CLINICAL TRIAL: NCT05555576
Title: Impact of Vitamin C on the Reduction of Opioid Consumption After an Emergency Department Visit for Acute Musculoskeletal Pain: A Double-Blind Randomized Control Trial Protocol
Brief Title: Impact of Vitamin C on opioïd Consumption After an Emergency Department Visit for Acute Musculoskeletal Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Raoul Daoust, Dr Emergency Medicine, Professor, Clinician Researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-2442
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Pain, Acute
Keywords: Vitamin C; Opioids; Emergency department; Pain
MeSH Terms: conditions — Acute Pain; Emergencies; Pain | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C (Experimental): 1 000 mg vitamin C taken orally twice a day
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1000 mg vitamin C taken orally twice a day (one in the morning and one in the evening) for a 14-day period after ED discharge for the treatment arm
  Arms: Vitamin C
Other: Placebo — Placebo taken orally twice a day (one in the morning and one in the evening) for a 14-day period after ED discharge for the treatment arm
  Arms: Placebo

SUMMARY:
Recent evidence has shown that vitamin C has some analgesic properties and can therefore reduce opioids used during healing. Vitamin C analgesic effect has been explored mostly during the short-term postoperative context or in disease specific chronic pain prevention but not after acute musculoskeletal injuries, which are often seen in the emergency department (ED).

The study's primary aim is to compare the total morphine 5 mg equivalent pills consumed during a two-week follow-up between patients receiving vitamin C or a placebo after ED discharge for an acute musculoskeletal pain complaint.

The investigators will conduct a double-blind randomized placebo-controlled trial with 464 participants distributed in two arms, one group receiving 1 000 mg of vitamin C twice a day for 14 days and another one receiving a placebo. Participants will be ≥18 years of age, treated in ED for acute musculoskeletal pain present for less than 2 weeks, and discharged with an opioid prescription for home pain management. Total morphine 5 mg equivalent pills consumed during the two-week follow-up will be assessed via an electronic (or paper) diary. In addition, patients will report their daily pain intensity, pain relief, side effects, and other types of pain medication or other non-pharmacological approach (ice, heat, immobilization, etc.) used. Three months after the injury, participants will also be contacted to evaluate chronic pain development. The investigators hypothesized that vitamin C, compared to a placebo, will reduce opioid consumption during a 14-day follow-up for ED discharged patients treated for acute pain.

DETAILED DESCRIPTION:
Study Rationale Literature suggests that the administration of vitamin C has an effect in reducing pain and opioid consumption in the context of immediate postoperative acute pain. However, the investigators could not find evidence on the effectiveness of vitamin C administration after an ED visit in the context of acute pain, notably in trauma injuries like fractures, bruises, sprains, strains, etc. Previous studies have only evaluated pain relief and opioid use for the immediate postoperative period of 24 to 72 hours. Therefore, the investigators propose to evaluate the efficacy of a 14-day regiment of vitamin C given to ED patients discharged with an opioid prescription for acute musculoskeletal (MSK) pain on total opioid consumption after two weeks. The two-week period was chosen because it defines the usual acute pain time frame, during which need for analgesics including opioids is essentially resolved in most patients (88% of our previous study cohort). Furthermore, since vitamin C is also associated with less post-herpetic neuralgia and complex regional pain syndromes (CRPS), the investigators also propose to evaluate its impact on the incidence of chronic pain and CRPS at 3 months.

Study Objectives The primary aim is to compare the difference in the total morphine 5 mg equivalent pills consumed after a two-week follow-up between patients receiving vitamin C versus patients receiving a placebo during these two weeks.

The secondary aims are to compare the following between patients receiving vitamin C vs patients receiving a placebo: pain intensity trajectories, average pain relief during the two-week, side effects, total morphine 5 mg equivalent pills consumed after a two-week follow-up for each type of MSK pain (fracture, contusions, cervical pain, lower back pain, MSK pain at other sites), incidence of chronic pain (including CRPS) at 3 months globally and for each type of MSK pain, incidence of CRPS for limb fractures, and for a wrist fracture in particular at 3 months, and prevalence of opioid use at 3 months.

Study Design The investigators will conduct a multi-center, double-blind, randomized, placebo-controlled trial performed in two tertiary trauma care university-affiliated hospitals located in Montreal and in Quebec City (Quebec, Canada) with an annual census of 60,000 and 67,000 visits, respectively.

Participants and recruitment Consecutive patients (from 8 to 20h every day) diagnosed with an acute musculoskeletal pain complaint ongoing for less than two weeks and discharged from the ED with an opioid prescription will be approached by the treating clinician to participate in the study and obtain their verbal consent to be seen by a research assistant. The decision to prescribe opioids will be at the discretion of the treating physician, but included patients will receive a standardized prescription of 20 pills of morphine 5 mg based on our previous work. The research assistant will then verify the patient's inclusion and exclusion criteria, explain the research protocol, and obtain informed written consent. Patients will be assessed via a two-week electronic (or paper) diary and contacted 3 months after ED discharge.

Randomization method and blinding Eligible patients will be block randomized at the initial visit (via 1:1 ratio) to either 1 000 mg vitamin C taken orally twice a day or matching placebo, using a centralized randomisation web system. Allocation concealment will be in place to ensure that the investigator and the individual enrolling the subject into the study have no prior knowledge of group assignment. Since fractures are associated with more opioid consumption, randomization will be a stratified by fracture or not and centre. According to the centralized web system, an independent pharmacist will dispense pre-packed numbered bottles of either vitamin C or placebo capsules for each patient. Both will be dispensed an identical capsules and the pharmacist will be unaware of the trial-group assignments. Each participant will be assigned a number and received the capsules in the corresponding pre-packed bottle. Group allocation will be disclosed only after final analysis or at the request of the patient's treating clinician.

Study drug Vitamin C (ascorbic acid) is a vital nutrient; it helps form and maintain bones, skin, and blood vessels and has antioxidant properties. It is not produced by the human body but occurs naturally in fruits and vegetables and other foods. It is also available as supplement over the counter in pharmacies, supermarkets, and health supplements stores and online. For adults, the recommended daily amount of vitamin C is 65 to 90 milligrams (mg) a day (Recommended Dietary Allowances by the Government of Canada).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and over;
2. Treated in ED for acute musculoskeletal pain present for less than 2 weeks;
3. Discharged with an opioid prescription;
4. Speaks French or English.

Exclusion Criteria:

1. Opioid use 1 month prior to the ED visit;
2. Already taking vitamin C supplement;
3. Active cancer;
4. Treated for chronic pain;
5. Treated for opioid use disorder;
6. Unable to fill out diary or unavailable for follow-up;
7. Any allergy, intolerance or sensitivity to milk (lactose) or morphine
8. Treated with cyclosporin or coumadin
9. Pregnant or lactating (dosage > 1,800 mg not recommended. For women of child-bearing age and sexually active in the past 3 months, a urine pregnancy test will be performed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in the total morphine 5 mg equivalent pills consumed | 14 days
  Compare the difference in the total morphine 5 mg equivalent pills consumed after a two-week follow-up between patients receiving vitamin C versus patients receiving a placebo during these two weeks.

SECONDARY OUTCOMES:
Pain intensity trajectories | 14 days
  Compare pain intensity trajectories, measured on an 11-point numerical rating scale (NRS) from 0 to 10 (0 is no pain and 10 worst pain imaginable), between both groups with group-based trajectory modelling.
Average pain relief | 14 days
  Patient's average pain relief during the two-week, measured on an 11-point numerical rating scale (NRS) from 0 to 10 (0 is no pain and 10 worst pain imaginable).
Number (%) of participants with side effects | 14 days
  Patients will report which of the following side effects were experienced during the 14-day period: nausea, vomiting, constipation, dizziness, drowsiness, sweating, weakness, or other side effects.
Total morphine 5 mg equivalent pills consumed for each type of musculoskeletal (MSK) pain | 14 days
  Fracture, contusions, cervical pain, lower back pain, MSK pain at other sites
Incidence of chronic pain (including complex regional pain syndrome (CRPS)) globally and for each type of MSK pain | 3 months
  Globally and for each type of MSK pain using pain disability index (PDI) or Budapest criteria
Incidence of CRPS for limb fractures, and for a wrist fracture | 3 months
  For these cases in particular using Budapest criteria
Prevalence of opioid use | 3 months
  Patients will be asked if they still consumed opioids at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Daoust, MD MSc, Principal Investigator — Université de Montréal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daoust R, Paquet J, Williamson D, Huard V, Arbour C, Perry JJ, Emond M, Berthelot S, Archambault P, Rouleau D, Morris J, Cournoyer A. Impact of vitamin C on the reduction of opioid consumption for acute musculoskeletal pain: A double-blind randomized control pilot study. PLoS One. 2024 Dec 31;19(12):e0316450. doi: 10.1371/journal.pone.0316450. eCollection 2024. PMID 39739762
- [Derived] Daoust R, Paquet J, Chauny JM, Williamson D, Huard V, Arbour C, Emond M, Rouleau D, Cournoyer A. Impact of vitamin C on the reduction of opioid consumption after an emergency department visit for acute musculoskeletal pain: a double-blind randomised control trial protocol. BMJ Open. 2023 May 24;13(5):e069230. doi: 10.1136/bmjopen-2022-069230. PMID 37225265